CLINICAL TRIAL: NCT00619307
Title: A Randomized, Multicenter, Two-arm, Open-label, Phase IIIb Study to Evaluate the Satisfaction in Relapsing Multiple Sclerosis Subjects Transitioning to Rebif® New Formulation From Rebif® (Interferon Beta-1a) With Ibuprofen When Necessary (PRN) or as Prophylaxis
Brief Title: Transition to Rebif New Formulation
Acronym: TRANSFER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 27571
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Results first posted 2010-07-26 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — Ibuprofen

ARMS (2):
- Transition with prophylactic ibuprofen (Active Comparator)
  Interventions: Drug: Rebif New Formulation + prophylactic Ibuprofen
- Transition with PRN ibuprofen (Active Comparator)
  Interventions: Drug: Rebif New Formulation + ibuprofen PRN

INTERVENTIONS:
Drug: Rebif New Formulation + prophylactic Ibuprofen — Subjects, currently on Rebif® 44 mcg three times a week, using Rebiject II as an injection device and having received Rebif® full dose 44 mcg three times a week for at least 6 months, receives systematically 400 mg ibuprofen as prophylactic treatment against flu-like symptoms on days when Rebif New Formulation 44 mcg three times a week is injected
  Arms: Transition with prophylactic ibuprofen
Drug: Rebif New Formulation + ibuprofen PRN — Subjects, currently on Rebif® 44 mcg three times a week, using Rebiject II as an injection device and having received Rebif® full dose 44 mcg three times a week for at least 6 months, should not administer Ibuprofen before the first Rebif New Formulation injection. If flu-like symptoms occur after the 44 mcg Rebif New Formulation injection then the subject can administer 400 mg ibuprofen. This should only be administered after the Rebif New Formulation injection and not before the Rebif New Formulation injection.
  Arms: Transition with PRN ibuprofen

SUMMARY:
To assess patient satisfaction with respect to the incidence of flu-like symptoms (FLS) in patients with multiple sclerosis transitioned from current Rebif (subcutaneously injected interferon beta-1a, 44 mcg three-times-weekly) to the new formulation of Rebif (RNF) while receiving ibuprofen either prophylactically or only when necessary (PRN) after the occurence of flu-like symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subject with relapsing forms of Multiple Sclerosis (MS)
* Expanded disability status scale (EDSS) score < 5.5 at study entry
* Subjects who have been administering Rebif 44 mcg three times a week for at least 6 months prior to study enrolment
* Subject currently using Rebiject II and who will use their own Rebiject II for the Rebif New Formulation injections
* Subject is between 18 and 60 years old inclusive
* Female subjects must be neither pregnant nor breast-feeding and must lack childbearing potential, as defined by either: post-menopausal or surgically sterile, or use a highly effective method of contraception.
* Subject is willing to follow study procedures
* Subject is willing and must not present any contra-indication to taking ibuprofen during 4 weeks of the study
* Subject has given written informed consent

Exclusion Criteria:

* Secondary Progressive Multiple Sclerosis without superimposed attacks
* Use of any other injectible medications during the week prior to the screening period, during the screening or treatment periods
* Subject receiving MS therapy in addition (i.e. combination therapy) to Rebif within 3 months prior to study enrolment or at any time during study protocol
* History of any chronic pain syndrome
* Subjects that use any investigational drug or experimental procedure within 12 weeks of visit
* Subject received corticosteroids or adrenocorticotrophic hormone (ACTH) within 30 days of visit 1
* Subject with flu-like symptoms (FLS) associated with any cause (i.e. no current flu and no FLS related to Interferon in the week prior to baseline)
* Subject has abnormal liver function, defined by a total bilirubin > 1.5 times the upper limit of normal, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 times the upper limit of the normal values.
* Subject has inadequate bone marrow reserve, defined as a total white blood cell count < 3.0 x 109/L, platelet count < 75 x 109/L, haemoglobin < 100 g/L.
* Subject suffers from an active autoimmune disease other than MS
* Subject suffers from major medical or psychiatric illness
* Subject has seizures history or is currently experiencing seizures not adequately controlled by anti-epileptics
* Subject is pregnant or attempting to conceive
* Visual or physical impairment that precludes completion of diaries and questionnaires by himself/herself
* Contraindication to ibuprofen:known hypersensitivity to the active ingredient ibuprofen
* Known hypersensitivity to non-steroidal anti-inflammatory drugs which can lead to asthmatic attacks, gastric and/or intestinal ulcers, gastro-intestinal bleeding, cerebro-vascular bleeding or other active bleeding, severe hepatic dysfunction, severe kidney dysfunction, severe cardiac insufficiency, or systemic lupus erythematosus

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Latour, MD, Study Director — Merck Serono International S.A., an affiliate of Merck KGaA, Darmstadt, Germany
Locations (2):
- Local Medical Information, Paris, France
- Local Medical Information, Munich, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 16 July 2007 and attended the last visit on 11 April 2008. One hundred and twenty three subjects gave informed consent and 117 were enrolled. Of these, all were treated except one subject scheduled to receive prophylactic ibuprofen, who withdrew consent before treatment.
Pre-assignment Details: There were 17 active centres, 6 centres in France and 11 centres in Germany. Screening visit took place within 2 weeks of randomisation. Six subjects were screening failures.
Groups:
- Transition With Prophylactic Ibuprofen: subjects received ibuprofen as prophylactic treatment against FLS on days when RNF 44 mcg tiw was injected (3 times weekly). Mandatory 400 mg of ibuprofen was administered prophylactically 30 to 60 minutes before each RNF injection.
  Optionally the subject could take another 400 mg 6 hours after the first ibuprofen dose or upon waking if more than 6 hours later and if necessary a third dose of 400 mg 6 hours later, adding up to a maximum of 1200 mg within 24 hours.
- Transition With PRN Ibuprofen: subjects were instructed not to administer ibuprofen before the first RNF injection. Ibuprofen was taken solely as needed, PRN, after RNF injections to alleviate the symptoms of FLS. If FLS occurred after a RNF injection, then the subject could administer the first dose of ibuprofen 400 mg. The second dose of ibuprofen 400 mg could be taken 6 hours after the first ibuprofen dose or upon waking if more than 6 hours later and if necessary a third dose of 400 mg 6 hours later, adding up to a maximum of 1200 mg within 24 hours of RNF injection.
Period: Overall Study
Arm/Group | Transition With Prophylactic Ibuprofen | Transition With PRN Ibuprofen
Started | 60 | 57
Completed | 56 | 53
Not Completed | 4 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrew consent | 1 | 0
Not completed — Severe migraine | 0 | 1
Not completed — MS attack plus steroids | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transition With Prophylactic Ibuprofen | Transition With PRN Ibuprofen | Total
Number analyzed (Participants) | 60 | 57 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 57 | 117
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (8.4) | 41.5 (8.9) | 41.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 40 | 88
  Male | 12 | 17 | 29
Region of Enrollment [Number; unit: participants]
  France | 14 | 14 | 28
  Germany | 46 | 43 | 89

OUTCOME MEASURES:

1. Primary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Flu-like Symptom Score
Description: This is defined as the sum of the scores for the "side effects" section questions 1-4, with a minimum possible total score of 1 and a maximum possible total score of 20 in the MSTCQ. The lower the score, the better the outcome.
Time Frame: 4 weeks
Population: ITT
Measure: Mean (95% Confidence Interval); unit: MSTCQ score (units on a scale)
Arm/Group | Transition With Prophylactic Ibuprofen | Transition With PRN Ibuprofen
Number analyzed (Participants) | 56 | 54
MSTCQ score (units on a scale) | 8.5 [7.4 to 9.6] | 9.1 [8.1 to 10.2]

2. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Total Score
Description: This is defined as the sum of the scores for the "injection systems" section questions 1-9 and the "side effects" section questions 1-11, with a minimum possible total score of 20 and a maximum possible total score of 100. The lower the score, the better the outcome.
Time Frame: 4 weeks
Population: ITT
Measure: Mean (95% Confidence Interval); unit: MSTCQ score (units on a scale)
Arm/Group | Transition With Prophylactic Ibuprofen | Transition With PRN Ibuprofen
Number analyzed (Participants) | 57 | 54
MSTCQ score (units on a scale) | 36.8 [34.5 to 39.1] | 38.3 [35.4 to 41.1]

3. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Injection Satisfaction Score
Description: This is defined as the sum of the scores for the "injection systems" section questions 1-9, with a minimum possible total score of 9 and a maximum possible total score of 45. The lower the score, the better the outcome.
Time Frame: 4 weeks
Population: ITT
Measure: Mean (95% Confidence Interval); unit: MSTCQ score (units on a scale)
Arm/Group | Transition With Prophylactic Ibuprofen | Transition With PRN Ibuprofen
Number analyzed (Participants) | 57 | 55
MSTCQ score (units on a scale) | 14.3 [13.3 to 15.2] | 15.0 [13.8 to 16.1]

4. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Injection Site Reaction Score
Description: This is defined as the sum of the scores for the "side effects" section questions 5 to 8, with a minimum possible total score of 1 and a maximum possible total score of 20. The lower the score, the better the outcome.
Time Frame: 4 weeks
Population: ITT
Measure: Mean (95% Confidence Interval); unit: MSTCQ score (units on a scale)
Arm/Group | Transition With Prophylactic Ibuprofen | Transition With PRN Ibuprofen
Number analyzed (Participants) | 57 | 54
MSTCQ score (units on a scale) | 9.4 [8.5 to 10.3] | 9.2 [8.0 to 10.4]

5. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Global Side Effects Score
Description: This is defined as the sum of the scores for "side effects" section questions 9 to 11, corresponding to minimum possible total score of 3 and a maximum possible total score of 15. The lower the score, the better the outcome.
Time Frame: 4 weeks
Population: ITT
Measure: Mean (95% Confidence Interval); unit: MSTCQ score (units on a scale)
Arm/Group | Transition With Prophylactic Ibuprofen | Transition With PRN Ibuprofen
Number analyzed (Participants) | 57 | 55
MSTCQ score (units on a scale) | 4.7 [4.2 to 5.1] | 5.0 [4.4 to 5.6]

ADVERSE EVENTS:
Time Frame: 4 Weeks
Description: Each subject was given a diary card for recording any adverse events. The table of Other Adverse Events shows all adverse events occurring at or above the reporting threshold.
Arm/Group | Transition With Prophylactic Ibuprofen | Transition With PRN Ibuprofen
Serious Adverse Events (participants affected / at risk) | 1/59 | 0/57
Other Adverse Events (participants affected / at risk) | 50/59 | 47/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transition With Prophylactic Ibuprofen (N=59) | Transition With PRN Ibuprofen (N=57)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transition With Prophylactic Ibuprofen (N=59) | Transition With PRN Ibuprofen (N=57)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 3 (3)
Chills (General disorders) | 4 (5) | 4 (5)
Fatigue (General disorders) | 15 (36) | 7 (10)
Influenza-like illness (General disorders) | 39 (182) | 38 (170)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (17)
Headache (Nervous system disorders) | 22 (41) | 16 (33)
Migraine (Nervous system disorders) | 0 (0) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other